CLINICAL TRIAL: NCT04017338
Title: Transplantation Using Hepatitis C Positive Donors to Hepatitis C Negative Recipients: A Safety Trial
Brief Title: Transplantation Using Hepatitis C Positive Donors, A Safety Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jordan Feld (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor-Investigator, Jordan Feld, Hepatologist and Senior Scientist, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JF-8-2018
Record Dates: First submitted 2019-07-02; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Lung Transplant Infection; Heart Transplant Infection; Kidney Transplant Infection; Kidney Pancreas Infection; Hepatitis C
Keywords: Organ Transplant; Hepatitis C Virus; Direct-Acting Antivirals (DAAs)
MeSH Terms: conditions — Hepatitis C | interventions — glecaprevir; pibrentasvir; Tablets; Ezetimibe

STUDY DESIGN:
Intervention Model Description: Investigators aim to transplant 40 recipients (20 lung; 20 other organs) on the transplant wait-list. Donor organs will be selected based on usual donor selection criteria. Recipients will be selected based on usual hospital protocol for selecting suitable recipients. After transplantation, recipients will receive highly effective antiviral prophylaxis using approved direct-acting antivirals (DAAs) Glecaprevir/Pibrentasvir (G/P) and they will also receive ezetimibe, a cholesterol-lowering medication. Additionally, lung transplant recipients will receive donor lungs treated with normothermic ex vivo lung perfusion (EVLP) prior to transplant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non Randomized Intervention (Experimental): Intervention description: recipients on the wait-list for lung, heart, kidney, and/or pancreas transplants will all receive antiviral treatment in the form of 8 total doses of oral tablets. Lung recipients will also receive donor lungs that are treated with normothermic EVLP (details of both described below).
  Drug: All recipients will receive glecaprevir (300mg)/pibrentasvir (120mg) supplied as three tablets per dose 6-12 hours prior to transplant, and for 7 days post-transplant. Other Names: Maviret. Patients will also receive ezetimibe (10mg), supplied as one tablet per dose to be taken at the same time as Maviret tablets (6-12 hours prior to transplant in addition to 7 daily doses post-transplant).
  Ex Vivo Lung Perfusion (EVLP): Normothermic EVLP is a method of donor lung preservation, assessment, treatment, and repair of injured organs. This method allows donor lungs to be treated for at least 12h under protective physiological conditions. Other names: Normothermic EVLP.
  Interventions: Drug: Glecaprevir 300 MG / Pibrentasvir 120 MG Oral Tablet; Drug: Ezetimibe 10Mg Oral Tablet; Device: Ex Vivo Lung Perfusion

INTERVENTIONS:
Drug: Glecaprevir 300 MG / Pibrentasvir 120 MG Oral Tablet — A potent and effective antiviral medication that has recently been approved for use in Canada with over 99% cure rates.
  Other Names: Maviret
Drug: Ezetimibe 10Mg Oral Tablet — A cholesterol-lowering medication that also blocks entry of HCV into liver cells.
Device: Ex Vivo Lung Perfusion — A technology that allows for the assessment and treatment of lungs prior to transplant.
  Other Names: Normothermic EVLP

SUMMARY:
The success of transplantation is significantly hindered by the lack of sufficient number of available donors. Many potential donor organs cannot be utilized in clinical transplantation because donors have chronic viral infections such as hepatitis C (HCV) infection. This study will test the possibility of safely transplanting organs from HCV-infected donors into HCV-uninfected recipients. Prior to transplantation, recipients will receive an initial dose of highly effective antiviral prophylaxis using approved direct-acting antivirals (DAAs) Glecaprevir/Pibrentasvir (G/P) and they will also receive ezetimibe, a cholesterol-lowering medication that also blocks entry of HCV into liver cells. They will then receive daily dosing of the same medications for 7 days after transplant. The aim of the study is to show that transplantation of organs from HCV+ donors is safe in the era of DAAs. The investigators hypothesize that rates of HCV transmission to recipients will be prevented by the use of DAA prophylaxis and any HCV transmission that does occur will be readily treatable and curable. If successful, the knowledge from this study can have a large impact to patients with end stage organ diseases by providing a large novel source of donors for organ transplantations.

DETAILED DESCRIPTION:
The investigators aim to transplant 40 recipients with end-stage organ disease (20 lung, and 20 other organs) using organs from HCV+ donors. Lungs to be used for transplantation will be exposed to ex vivo lung perfusion with use of ultraviolet C light during perfusion if clinically indicated for lung-related outcomes (ie. not determined by the study investigators). Ex vivo organ perfusion will not be used for other organs. Recipients who are scheduled to receive an HCV-infected organ will receive glecaprevir (300mg)/pibrentasvir (120mg) supplied as three fixed-dose combination tablets once a day starting prior to the transplant as soon the patient is in the hospital and it is confirmed that the transplant is proceeding. HCV treatment will continue for 7 days post-transplant (total 8 doses). Recipients will also receive ezetimibe (10 mg) once daily starting at the same time as G/P and continued until 7 days post-transplant. Recipients will have blood samples taken daily for the first 2 weeks and then weekly until 12 weeks post-transplant for HCV PCR (with additional final sample taken at 6 months post-transplant). The investigators hypothesize that HCV transmission to recipients will be prevented by the use of potent DAA prophylaxis plus ezetimibe with or without ex vivo organ perfusion in the immediate peri-operative period.

ELIGIBILITY:
Donor Inclusion Criteria:

* Age <70
* NAT+ HCV donor

Donor Exclusion Criteria:

* HIV positive or HTLV 1/2 positive
* Hepatitis B surface Antigen positive
* Any medical issues in the donor that would normally clinically exclude the donor (e.g. history of cancer, evidence of organ dysfunction, etc)
* Age>70

Recipient Inclusion Criteria:

* Recipients listed for kidney, kidney-pancreas, pancreas transplant alone, heart, or lung transplant
* HCV NAT negative
* Provides written informed consent

Recipient Exclusion Criteria:

* Chronic liver disease with > stage 2 fibrosis
* Participating in another interventional clinical trial
* Recipient listed for liver transplant
* Known allergy or contraindication to Glecaprevir/Pibrentasvir or ezetimibe

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-transplant Survival [Safety] | 6 months
  Survival at 6 months post-transplantation in patients receiving organs from HCV-positive donors reported as a binary variable (survival: yes vs. no).
Incidence of HCV transmission [Safety] | 6 months
  Incidence of HCV transmission following organ transplantation using HCV-positive donors. The proportion who are HCV RNA positive by PCR at 6 months post-transplantation will be reported as a binary variable (transmission: yes vs. no).
Incidence of treatment-emergent adverse events [Safety and Tolerability] | 30 days
  The number and type of adverse events that are related to treatment with glecaprevir/pibrentasvir or ezetimibe in the opinion of the investigator will be reported at 30 days.

SECONDARY OUTCOMES:
Long-Term Organ Function using Spirometry for Lung Recipients | 1 year
  Spirometry (also known as a pulmonary function test) will be used to assess lung function, measured as the Forced Vital Capacity (FVC) in liters.
Long-Term Organ Function using Exercise Tolerance for Lung Recipients | 1 year
  A 6-minute walk test will also be used to assess lung function, measured as the total distance the patient can walk during the span of 6 minutes in meters).
Long-Term Organ Function for Pancreas Recipients | 1 year
  Insulin dependency will be used to assess pancreas function in patients with diabetes, measured as the status of insulin freedom (not needing insulin) after the first year post transplantation. The outcome will be reported as a binary variable (insulin freedom: yes vs. no).
Long-Term Organ Function for Kidney Recipients | 1 year
  Creatinine levels will be used to assess kidney function and will be collected with a blood test. The estimated glomerular filtration rate (eGFR) will then be calculated in milliliters per minute using serum creatinine (Scr). The formula used to calculate eGFR will be using the Modification of Diet in Renal Disease (MDRD) equation, GFR (mL/min/1.73 m2) = 175 x (Scr)-1.154 x (Age)-0.203 x (0.742 if female) x (1.212 if African American)
Long-Term Organ Function for Heart Recipients | 1 year
  Left ventricular ejection fraction (the amount of blood leaving the heart during each contraction) will be measured by echocardiography and will be expressed as a percentage.
Acute Cellular Rejection | 1 year
  The incidence of acute cellular rejection following transplantation will be measured as the proportion of patients with biopsy-proven acute cellular rejection of the transplanted organ and will be reported as a binary variable (yes vs. no).
HCV Seroconversion | 1 year
  HCV seroconversion will be measured as the proportion of patients who test positive for antibodies to HCV at 1 year post-transplant and will be reported as a binary variable (HCV antibody positive: yes vs. no)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Feld, MD, MPH, Principal Investigator — University Health Network Toronto General Hospital
Locations (1):
- University Health Network Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feld JJ, Cypel M, Kumar D, Dahari H, Pinto Ribeiro RV, Marks N, Kamkar N, Bahinskaya I, Onofrio FQ, Zahoor MA, Cerrochi O, Tinckam K, Kim SJ, Schiff J, Reichman TW, McDonald M, Alba C, Waddell TK, Sapisochin G, Selzner M, Keshavjee S, Janssen HLA, Hansen BE, Singer LG, Humar A. Short-course, direct-acting antivirals and ezetimibe to prevent HCV infection in recipients of organs from HCV-infected donors: a phase 3, single-centre, open-label study. Lancet Gastroenterol Hepatol. 2020 Jul;5(7):649-657. doi: 10.1016/S2468-1253(20)30081-9. Epub 2020 May 6. PMID 32389183